CLINICAL TRIAL: NCT03486925
Title: An Eye-tracking Study to Investigate Oxytocin Effect on Attention Inhibition
Brief Title: Oxytocin Effect on Attention Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: UESTC-neuSCAN-45
Record Dates: First submitted 2018-03-27; First posted 2018-04-03 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Healthy
Keywords: oxytocin, eye-tracking, attention inhibition

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- oxytocin group (Experimental)
  Interventions: Drug: oxytocin treatment
- placebo group (Placebo Comparator)
  Interventions: Drug: placebo treatment

INTERVENTIONS:
Drug: oxytocin treatment — intranasal administration of oxytocin (24IU)
  Arms: oxytocin group
Drug: placebo treatment — intranasal administration of placebo
  Arms: placebo group

SUMMARY:
Effects of intranasal oxytocin (24IU) on cognitive control of attention

DETAILED DESCRIPTION:
The cognitive control of attention towards neutral and emotional stimuli represents a key functional domain and disruptions in this domain have been associated with a range of psychiatric disorders. Saccadic eye movement tasks have been used to assess individual differences in the cognitive control of attention and alterations in psychiatric disorders. Recent evidence suggests that the hypothalamic neuropeptide Oxytocin (OXT) may modulate attention allocation and regulation. To this end the present randomized between-subject placebo-controlled experiment examined whether intranasal OXT modulates behavior in an eye-tracking saccade / anti-saccade paradigm in healthy male subjects. The paradigm used non-social (neutral shape) as well as social (happy, sad, angry, fear, and neutral faces) stimuli to explore emotion-specific effects of OXT.

ELIGIBILITY:
Inclusion Criteria:

* Male, healthy participants
* Non smokers

Exclusion Criteria:

* Previous or current medical, psychiatric, neurological disorder
* Regular medication
* Use of any psychoactive substances in the 24 hours before experiment
* Contra-indications for oxytocin
* Contra-indications for eye-tracking data acquisition

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2017-12-19 (Actual); Primary Completion 2018-07-20 (Actual); Study Completion 2018-08-28 (Actual)

PRIMARY OUTCOMES:
emotion-specific saccade latencies | 45 minutes - 100 minutes after treatment
  comparison between emotion-specific saccade latencies between the treatment groups (in milliseconds)
emotion-specific error rates | 45 minutes - 100 minutes after treatment
  comparison between the emotion-specific ratio of unsuccessful anti-saccades between the treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- School of Life Science and Technology, University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No